CLINICAL TRIAL: NCT02060019
Title: A Phase I Clinical Trial to Investigate the Pharmacokinetic Interactions and Safety Between Exforge Tab. and Crestor Tab. in Healthy Male Subjects
Brief Title: Pharmacokinetic Interactions and Safety Between Exforge Tab. and Crestor Tab. in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: CJ_EXR_101
Record Dates: First submitted 2014-02-06; First posted 2014-02-11 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy
Keywords: Pharmacokinetics; Pharmacodynamics; Safety; Tolerability
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- exforge 10/160mg(amlodipine 10mg, valsartan160mg) (Experimental): 1 tablet daily for 10days
  Interventions: Drug: administration of exforge 10/160mg for 3days. Next 7days administration of exforge 10/160mg and crestor 20mg.
- crestor 20mg(rosuvastatin 20mg) (Experimental): 1 tablet daily for 7days
  Interventions: Drug: administration of exforge 10/160mg for 3days. Next 7days administration of exforge 10/160mg and crestor 20mg.

INTERVENTIONS:
Drug: administration of exforge 10/160mg for 3days. Next 7days administration of exforge 10/160mg and crestor 20mg.

SUMMARY:
This study is designated to evaluate the pharmacokinetic interactions of amlodipine besylate, valsartan and rosuvastatin in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Male volunteers in the age between 20 and 55 years old
2. The weight range is not exceed ±20% of ideal weight Ideal weight = [height -100]*0.9
3. Subjects with no history of any significant chronic disease
4. Judged to be in good health on the basis of their electrocardiography (ECG) and routine laboratory data obtained within 3 weeks prior to study drug administration
5. Willing to adhere to protocol requirements and sign a informed consent form

Exclusion Criteria:

1. History of clinically significant allergies including drug allergies
2. History of clinically significant hepatic, renal, gastrointestinal, pulmonary, ,musculoskeletal, endocrine, psychiatric, hematologic, oncologic, neurologic or cardiovascular disease
3. History of genetic muscular disease and family history
4. hypotension (Systolic Blood Pressure(SBP) ≤ 105 or Diastolic Blood Pressure(DBP) ≤ 65) or hypertension(SBP ≥ 150 or DBP ≥ 100)
5. AST(Aspartate Transaminase), ALT(ALanine Transaminase), total bilirubin( > 1.5 times to normal range
6. Creatinine clearance < 80mL/min
7. Subjects with a history of gastrointestinal diseases which might significantly change ADME(Absorption, Distribution, Metabolism and Excretion) of medicines
8. Serious injury, surgery and acute illness within 4 weeks prior to drug administration
9. History of alcohol, smoking abuse

   * alcohol > 21 units/week, 1 unit=10g=12.5mL of pure alcohol
   * smoking > 10 cigarettes/day
10. Use of any other medication, including herbal products, within the 2 weeks before dosing
11. Participated in a previous clinical trial within 3 months prior to drug administration
12. Subjects with whole blood donation within 2 months, component blood donation within months prior to drug administration
13. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
14. Clinical laboratory test values are positive (HBsAg, HCV Ab, HIV Ag/Ab, VDRL)
15. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2014-03; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Assessment of the drug-drug interactions of amlodipine, valsartan and rosuvastatin: Cmax,ss(Maximum steady-state plasma drug concentration during a dosage interval ), AUCτ(Area Under the Curve) | 3 days
  after steady state (Administration of Investigational Product 7day or 10days)

SECONDARY OUTCOMES:
Assessment of the amlodipine, valsartan and rosuvastatin : AUCinf, tmax,ss(Time to reach Cmax,ss), t1/2 | 3 days
  steady state (Administration of Investigational Product)

CONTACTS AND LOCATIONS:
Overall Officials: Young Ran Yoon PhD, Principal Investigator — Kyungpook university hostipal
Locations (1):
- Kyungpook university hospital, Deagu, South Korea